CLINICAL TRIAL: NCT04829045
Title: The Effect of Acupuncture as Adjunctive Therapy on Homeostasis Model Assessment-insulin Resistance and Health Related Quality of Life in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Acupuncture as Adjunctive Therapy in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Cheok Yean Chin, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT04829045; JKEUPM-2018-294 (Other: JKEUPM of Universiti Putra Malaysia); U1111-1219-3545 (Other: Universal Trial number)
Record Dates: First submitted 2020-12-23; First posted 2021-04-02 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2; Acupuncture
Keywords: Type 2 diabetes mellitus; Acupuncture; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture plus diabetic routine care (Experimental): Subjects will receive acupuncture treatment using press needles
  Interventions: Device: SEIRIN PYONEX Acupuncture Needles
- Placebo plus diabetic routine care (Placebo Comparator): Subjects are given placebo
  Interventions: Other: PYONEX Placebo

INTERVENTIONS:
Device: SEIRIN PYONEX Acupuncture Needles — 10 press needles (PYONEX ø0.20×1.5mm made by Seirin Corporation) will be placed on abdomen area; 10 sessions over 6 weeks.
  Arms: Acupuncture plus diabetic routine care
Other: PYONEX Placebo — Subjects are given placebo on abdomen area; 10 sessions over 6 weeks.
  Arms: Placebo plus diabetic routine care

SUMMARY:
This study aims to determine the effect of acupuncture as an adjunctive therapy on homeostasis model assessment-insulin resistance (HOMA-IR) and health-related quality of life (HRQoL) in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo controlled and parallel design trial. Participants will be randomized to either acupuncture (n=30) or placebo (n=30) using a 1:1 ratio. The permuted blocks with a block size of 2 will be used. Both groups will continue with their routine diabetes care. Primary outcome of HOMA-IR will be measured at the time of recruitment (baseline) and after completion of 10 sessions (week 7) of the treatment. Secondary outcome of HRQOL will be measured at the time of recruitment (baseline), after completion of 5 sessions (week 3/4) and 10 sessions (week 7) of the treatment while outcomes of body mass index and waist circumference are measured at the time of recruitment (baseline) and after completion of 10 sessions (week 7) of the treatment. Any adverse event will be recorded at every visit. The sequence generation and allocation will remain concealed from the patient and practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose (FPG) ≥ 7.0 mmol/L [126 mg/dL] or HbA1c ≥ 6.5%.
* Subjects have had type 2 diabetes mellitus for more than one year
* Receive oral anti-diabetic agents on a stable dose over the previous 3 months.

Exclusion Criteria:

* Under insulin therapy
* With other acute or chronic health problems
* Body mass index (BMI) ≥ 40.0 kg/m²
* Needle phobia or allergy to adhesive plaster
* Planning to move out from Malaysia within 4 months'
* Being pregnant, planning for pregnancy or lactating women

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fasting serum insulin | change from baseline fasting serum insulin at 7 weeks
  Analyzed in μU/ml using heparin tube
Fasting plasma glucose | change from baseline fasting plasma glucose at 7 weeks
  Analyzed in mmol l-^1 using sodium fluoride tube
Homeostasis model assessment- insulin resistance (HOMA-IR) | change from baseline HOMA-IR at 7 weeks
  Fasting serum insulin and fasting plasma glucose will be combined to report HOMA-IR in unit [fasting serum insulin (μU/ml)×fasting plasma glucose (mmol l-1)/22.5](Mathews et al., 1985).

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | change from baseline HRQoL at 3-4 weeks
  Changes is assessed using World Health Organization Quality of Life Assessment: Brief Version (WHOQoL-BREF [English/Malay]) questionnaire which consists of 26 items and the scores range from 0-100. The higher the score, the better the HRQoL.
Health-related quality of life (HRQoL) | change from baseline HRQoL at 7 weeks
  Changes is assessed using World Health Organization Quality of Life Assessment: Brief Version (WHOQoL-BREF [English/Malay]) questionnaire which consists of 26 items and the scores range from 0-100. The higher the score, the better the HRQoL.
Weight | change from baseline weight at 7 weeks
  Changes is measured using digital scale TANITA weighing machine in kilograms.
Body mass index | change from baseline body mass index at 7 weeks
  Weight and height will be combined to report BMI in kg/m^2. Height will be measured in centimeter using SECA body meter while weight will be measured in kilograms using digital scale TANITA weighing machine
Waist circumference | change from baseline waist circumference at 7 weeks
  Changes is measured using SECA measuring tape in centimeter
Incident of treatment adverse events in terms of intensity (grades 1 - 5) | 7 weeks
  Evaluated according to National Cancer Institute (2017) guidelines in terms of intensity (grade 1 - 5). Higher grades mean worst adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Cheok Yean Chin, MSc, OMBAcC, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheok YC, Mohd Shariff Z, Chan YM, Ng OC, Lee PY. Effectiveness of acupuncture as adjunctive therapy in type 2 diabetic: Study protocol for a randomized controlled trial. PLoS One. 2023 Sep 20;18(9):e0284337. doi: 10.1371/journal.pone.0284337. eCollection 2023. PMID 37729132